CLINICAL TRIAL: NCT05356481
Title: Comparison Of Segmental Vibration On Flexors and Extensor Muscle Groups On Upper Limb Function In Post-Stroke Patients
Brief Title: Effect of Segmental Muscle Vibration on Upper Limb Function in Post Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/01390 Shahid Shabbir
Record Dates: First submitted 2022-04-28; First posted 2022-05-02 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Stroke
Keywords: segmental muscle vibration,spasticity,upper limb function
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Assignment
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group A (Experimental): will recieve (low frequency segmental muscle vibration of 41 Hz over flexors muscles of upper limb Pectoralis minor, Biceps brachii, Flexor carpi muscle + general physical therapy session ) The transducer applied perpendicular to the muscle near its distal tendon insertion.The application consisted of 3 vibration sessions each with duration of 5 minutes for each muscle with 1 minute interval separated these sessions during the interval muscle vibration will interrupted and the subject will request to relax the muscle
  Interventions: Device: segmental muscle vibration
- Experimental Group B (Experimental): group receive (low frequency segmental muscle vibration of 41 Hz over extensors muscles of upper limb Triceps brachii, Extensor carpi radialis longus & brevis + general physical therapy session ) The transducer applied perpendicular to the muscle near its distal tendon insertion The application consisted of 3 vibration sessions each with duration of 5 minutes for each muscle with 1 minute interval separated these sessions during the interval muscle vibration will interrupted and the subject will request to relax the muscle
  Interventions: Device: segmental muscle vibration

INTERVENTIONS:
Device: segmental muscle vibration — Segmental muscle vibration will delivered over the target muscles by means of vibrator with general physical therapy session
  Other Names: general physical therapy session

SUMMARY:
The aim of this study is to observe and to compare effects of segmental vibration on flexors versus extensor muscle groups on upper limb function in post-stroke patients. This study will be helpful in finding out that either low frequency segmental vibration on flexors muscle group is better in improving upper limb function or low frequency segmental vibration on extensor muscle group is more beneficent in improving upper limb function.

DETAILED DESCRIPTION:
Stroke is the leading cause of long-term disability and is often associated with persistent involvement of upper limbs.Several disturbances are the manifestation of UL impairments after stroke (i.e., muscle weakness, changes in muscle tone, joint disturbances, impaired motor control) . Muscular weakness and spasticity are most commonly observed in post stroke patients. There are many strategies are developed to improve functional status and to reduce spasticity pattern in post stroke patients. Among the different approaches to improve motor functions in post stroke patients, vibration therapy gives strong stimulatory effects in post paretic limb. Segmental muscle vibration (SMV) is a fairly new technique that has been used to improve motor function and inhibit spasticity in the hemiplegic upper extremity of patients following a stroke. In SMV, a vibratory stimulus is applied to a specific muscle tendon using a mechanical device unit.The aim of this study is to observe and to compare effects of segmental vibration on flexors versus extensor muscle groups on upper limb function in post-stroke patients. This study will be helpful in finding out that either low frequency segmental vibration on flexors muscle group is better in improving upper limb function or low frequency segmental vibration on extensor muscle group is more beneficent in improving upper limb function.

ELIGIBILITY:
Inclusion Criteria:

* Both genders
* Age: between 50-65 years.
* Spasticity 1-3 on MAS
* 3-6 months post stroke patients

Exclusion Criteria:

* Cardiovascular event (myocardial ischemia or infarction) occurring within 12 months,
* Use of any antispastic drug
* Pain from vibration
* Inflammatory osteoarticular diseases

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2023-01-15 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Wolf Motor Functional Test | 10 to 15 minutes
  WMFT is valid and reliable on assessing upper extremities motor function of stroke patients. The WFMT is a tool with high interrater reliability, internal consistency, test-retest reliability and adequate stability.
Modified Ashworth Scale | 4 to 5 minutes
  This scale measures resistance during passive soft-tissue stretching and is used as a simple measure of spasticity
Fugl Meyer Assessment | 10 minutes
  Fugl Meyer Assessment
Manual Muscle Testing | 8 to 10 minutes
  to check muscle strength
• Brunnstrom Stages of Stroke Recovery • Brunnstrom Stages of Stroke Recovery Brunnstrom Stages of Stroke Recovery | 5 to 10 minutes
  to check the stages of improvemnet

CONTACTS AND LOCATIONS:
Overall Officials: Aruba Saeed, PhD*, Study Chair — Riphah international university.pakistan
Locations (2):
- Pakistan (2):
  - Muhammad shahid shabbir, Rawalpindi, Punjab Province
  - Riphah International University, Rawalpindi, Punjab Province

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shabbir MS, Saeed A, Tariq S, Shabbir N, Nasir R, Riaz H. Effects of segmental muscle vibration on flexor and extensor groups of the upper limb in enhancing functional recovery after stroke: A randomized trial. J Bodyw Mov Ther. 2025 Dec;45:1-7. doi: 10.1016/j.jbmt.2025.07.019. Epub 2025 Jul 25. PMID 41316550